CLINICAL TRIAL: NCT05479838
Title: Evaluation of the Predictive Effect of Inflammatory Markers in Predicting the Occurrence of Post-PCI Nephrotoxicity in MI Patients Admitted to the Emergency Department.
Brief Title: Evaluation of the Predictive Effect of Inflammatory Markers in MI Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Mustafa Enes DEMİREL, Assist. Prof., Abant Izzet Baysal University
Other Study IDs: BAIBU-EM-MED-1
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; Nephropathy; Inflammation Mediators
MeSH Terms: conditions — Myocardial Infarction; Kidney Diseases | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ST Elevation MI: ST-segment in adjacent ≥2 leads Elevation ( ≥2 mm in precordial leads, ≥1 mm in extremity leads) or left bundle branch block, ischemic type chest pain lasting longer than 30 minutes, and two or more elevations of serum creatine kinase myocardial band and troponin levels will be used as diagnostic criteria for STEMI. Patients with ST-elevation on the ECG will be referred to as STEMI, non -STEMI with twice the troponin level despite the absence of ST elevation. Patients who do not have ST elevation on ECG and whose troponin values do not exceed the reference range, but who are diagnosed as USAP presenting with typical chest pain and undergoing coronary angiography will be included in the study.
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — Coronary angiography will be performed via the femoral or radial artery, and primary PCI will be performed using standard guide catheters, guide wires, balloon catheters, and stents according to current guidelines. All PCI interventions performed by invasive cardiologists. The primary PCI type and contrast amount will be decided by the medical team. All patients will be treated by administering non-ionic, monomeric, low-osmolar iodinated iohexol as an intravascular contrast agent .

SUMMARY:
Acute myocardial infarction (AMI), triggered by myocardial ischemia and reperfusion injury, is a disease with high morbidity and mortality, and there is a tendency for its incidence to increase at younger ages.

One of the most worrisome complications of primary percutaneous surgery is contrast-induced nephropathy, which is associated with increased mortality and morbidity in myocardial infarction after coronary interventions. In many studies, inflammatory markers, which are thought to give an idea about the development of contrast-related nephropathy, have been examined.

The transcription factor nuclear factor erythroid 2-related factor 2 (Nrf2) is a master regulator of cytoprotective protein expression driven by antioxidant response agents (AREs) and plays a decisive role in the regulation of oxidative defense and redox homeostasis in cells.

There are studies showing the role of Nrf2 in the pathogenesis of kidney damage in some studies.

Studies on the effect of Nrf2 level on contrast media nephropathy in patients with contrast media nephropathy (CIN) are limited in the literature.

This study also aimed to form a basis for the literature, which is a small number of studies, in later studies.

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI), triggered by myocardial ischemia and reperfusion injury, is a disease with high morbidity and mortality, and there is a tendency for its incidence to increase at younger ages.

One of the most worrisome complications of primary percutaneous surgery is contrast-induced nephropathy and acute renal failure, which is associated with increased mortality and morbidity in myocardial infarction after coronary interventions. In many studies, markers that are thought to give an idea about the development of contrast-associated nephropathy have been examined. Acute renal failure (ARF) refers to a sudden decrease in glomerular tissue. Glomerular filtration rate (GFR) causes creatinine accumulation in the body and decreased urine output for various reasons, causing serious complications. Apart from dysfunction during the acute phase, there is a significant risk for permanent tissue damage. Therefore, kidney function cannot be restored, leading to the development of chronic renal failure (CKD), a sustained decrease in GFR, and increased long-term mortality. Incomplete recovery can also lead to the onset or further deterioration of chronic renal failure. Clinically, apart from hemodialysis treatment, few effective methods can treat the formation and development of ARF. Therefore, there is still an urgent need for new targets or better treatment options to prevent ARF and promote adaptive repair after ARF occurs. To date, the molecular mechanism of ARF is unclear, but there is increasing evidence that ARF is directly related to oxidative stress. In some studies, there are studies showing the role of Transcription factor nuclear factor erythroid 2-related factor 2 (Nrf2) in the pathogenesis of kidney damage.

There is an increase in mortality and morbidity rates due to nephrotoxicity after percutaneous intervention after MI. Studies showing that Nrf2 level may have a protective effect in contrast media nephropathy in patients with contrast media nephropathy (CIN) are limited in the literature.

The transcription factor nuclear factor erythroid 2-related factor 2 (Nrf2) is a master regulator of cytoprotective protein expression driven by antioxidant response agents (AREs) and plays a decisive role in the regulation of oxidative defense and redox homeostasis in cells. Although there are studies examining the epidemiological, demographic and clinical characteristics of patients in our country, studies on the importance of inflammatory parameters and the mortality and morbidity of Nrf2 levels are not available in our country.

This study aimed to form the basis of the literature, which is a small number of studies, in later studies.

ELIGIBILITY:
Inclusion Criteria:

* Those diagnosed with STEMI

Exclusion Criteria:

* Under 18 years of age
* With other clinical diagnoses in ED
* Pregnancy
* Acute or chronic kidney failure
* Malignancy
* Active infection
* Rheumatoid Diseases
* If patient want leave study
* Mortality in 28 days

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included in the study will be followed up after the percutaneous intervention with routine controls. CIN identification; Renal dysfunction (a 0.3 mg/dl increase in absolute serum creatinine or at least 1.5-fold increase in basal creatinine) within 7 days of intravenous contrast administration and contrast nephropathy as recommended by the Journal of the American College of Cardiology will be defined. Diagnosis, treatment, follow-up and discharge of patients will proceed according to routine medical procedures. In this study, a different procedure related to diagnosis, treatment, follow-up and discharge will not be used.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-15 (Estimated); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Nuclear factor erythroid 2-related factor 2 levels | 30 minutes
  The blood taken from the patients into biochemistry tubes at the time of application will be centrifuged at 1500 g for 10 minutes after the clotting process is completed, and their serum will be separated and stored at -80 C until the working day. On the working day, samples will be thawed and Nrf2 levels will be measured using commercially available kits.
  Nuclear Factor Erythroid 2-Related Factor 2 (BtLab) Product Summary Size: 96T Sensitivity: 0.11ng/ml Detection range: 0.2-60ng/ml Sample type: Serum, plasma, cell culture supernates Reactive with: Human https://www.bt-laboratory.com/index.php/Shop/Index/productShijiheDetail/p_id/987/cate/kit.html

SECONDARY OUTCOMES:
Troponin | 30 minutes
  The blood taken from the patients into biochemistry tubes at the time of application will be centrifuged at 1500 g for 10 minutes after the clotting process is completed, and their serum will be separated and stored at -80 C until the working day. On the working day, samples will be thawed and Troponin levels will be measured using commercially available kits.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Enes DEMİREL, M.D., Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant Izzet University faculty of Medicine Department of Emercengy Medicine, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No